CLINICAL TRIAL: NCT02818907
Title: Evaluation of Survival Prognostic Factors for Patients With Exocrine Pancreatic Cancer Resectable or Potentially Resectable : a Multicentre Prospective Cohort
Brief Title: Evaluation of Survival Prognostic Factors for Patients With Exocrine Pancreatic Cancer Resectable or Potentially Resectable
Acronym: Pancreas-CGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Cancéropôle Grand-Est (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pancreas-CGE
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

ARMS (1):
- Additional biological samples (Other): Additional blood samples will be realized specifically to the study at baseline, after neoadjuvant chemotherapy (if applicable) and before surgery, 1 month after surgery and 1 month after the last adjuvant chemotherapy cycle.
  Peripheral blood mononuclear cell (PBMC), plasma and circulating tumor DNA and RNA will be collected.
  Tumor tissue will be collected during surgery.
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — blood and tumor tissue samples

SUMMARY:
This study aims to collect clinical, biological and quality of life data from patients with a borderline or resectable pancreatic cancer. It will collect information from the date of diagnosis along the therapeutic care of the patients, and a 3-years follow-up after the end of the treatment. The database will be updated at each patient's visit. Biological samples will include: tumor, and plasma. Epidemiological data will also be collected, whereas Quality of life will be assessed by the EORTC standard. The objectives of this database are to identify new biomarkers (genomic, immunologic, and epidemiologic) and promote high quality standard research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with exocrine resectable pancreatic adenocarcinoma or potentially resectable (that after neoadjuvant treatment are considered appropriate candidates for resection)
* Histologically or cytologically documented diagnosis of exocrine pancreatic adenocarcinoma
* Written informed consent obtained prior enrollment in the study

Exclusion Criteria:

* other types of pancreatic cancer, in particular endocrine tumor or acinar cells
* ampulloma
* metastatic disease
* other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer
* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study
* patient under guardianship, curator or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
disease-free survival according to the consensus DATECAN (Bonnetain F et al, European Journal of Cancer 2014) | date of first disease apparition [within 3 years after the enrollment of the last patient]
  DATECAN = Definition for the Assessment of Time-to-event Endpoints in CANcer trials

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Institut de cancérologie de Lorraine, Nancy
  - Centre Hospitalier Universitaire Robert Debré, Reims
  - Centre Paul Strauss, Strasbourg
  - CHU de Strasbourg - Hautepierre, Strasbourg